CLINICAL TRIAL: NCT02087397
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Into the Corpus Cavernous in Patients With Erectile Dysfunction.
Brief Title: Autologous Adipose-Derived Stromal Cells Delivered Into the Corpus Cavernous in Patients With Erectile Dysfunction
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-US-ED-001
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Erectile Dysfunction
Keywords: Stem Cell; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AD-SVF Cell Injection (Experimental)
  Interventions: Other: Liposuction; Biological: AD-SVF Cell Injection

INTERVENTIONS:
Other: Liposuction — Liposuction using aspiration syringe and tumescent local anesthesia
  Other Names: Lipoaspiration
Biological: AD-SVF Cell Injection — Stem cell implantation will be performed using direct injection into the Corpus Cavernosum with local anesthesia
  Other Names: Adipose derived Stromal Vascular Fraction Cell Injection

SUMMARY:
This will be an open-label, non-randomized, multi-center, patient sponsored study of Adipose-Derived Stromal Vascular Fraction cells (AD-SVF) implantation delivered into the corpus cavernous in patients with Erectile Dysfunction.

The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the disease pathology of patients with diagnosed Erectile Dysfunction.

DETAILED DESCRIPTION:
AD-SVF will be collected from the patient's adipose-derived tissue (body fat). Using local anesthesia, Liposuction will be performed to collect the adipose tissue specimen. The adipose tissue is then transferred to the laboratory for separation of the adipose tissue derived stem cells. In addition, peripheral blood will be collected for isolation of platelet rich plasma, which are then combined with the ASC's for direct injection to the Corpus Cavernosum (Penis).

ELIGIBILITY:
Inclusion Criteria

* Males Age 18 and 80 years.
* Penile arterial insufficiency and or venous leakage (doppler) at the time o inclusion: PSV <25 cm/sec, PSV >25 cm/sec, EDV>5cm/sec, RI<0,75.
* Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria

* Severe co-morbidities like cardiac insufficiency, congestive cardiac failure (NYHA ≥ III), malignancy, infection, sepsis and bed sores.
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will be evaluated by an expert as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or \ interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg or greater than 200mmHg
* Resting heart rate > 100 bpm;
* Active clinical infection within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Schramek's Grade | Baseline, 3 months, and 6 months
  Schramek's grading system- penile rigidity Grade 1 - No erection Grade 2 - Slight Tumescence Grade 3 - Full volume without rigidity Grade 4 - Sufficient for sexual intercourse Grade 5 - Full erection

SECONDARY OUTCOMES:
Change from Baseline of Penile Doppler | Baseline and 6 moths
Improvement in Phallometry Measures | Baseline, 3 Months, and 6 Months
  Air Chamber Measurements/ Circumference Measurements

OTHER OUTCOMES:
Number of Participants with Adverse Events | Baseline, 3 Months, and 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khera M, Albersen M, Mulhall JP. Mesenchymal stem cell therapy for the treatment of erectile dysfunction. J Sex Med. 2015 May;12(5):1105-6. doi: 10.1111/jsm.12871. No abstract available. PMID 25974235